CLINICAL TRIAL: NCT01570023
Title: Comparison Between Isometric Lingual Strengthening Exercises and Standard Clinical Care for the Treatment of Dysphagia
Brief Title: Study of Tongue Strengthening for Swallowing Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0518
Record Dates: First submitted 2012-03-27; First posted 2012-04-04 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Dysphagia
Keywords: Deglutition; Exercise
MeSH Terms: conditions — Deglutition Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Clinical Care (No Intervention): Standard swallowing intervention is that which is identified by the SLP as appropriate to treat the patient's dysphagia and is in common clinical practice. Such treatment would consist of dietary or postural compensatory strategies (i.e., chin down posture while swallowing).
- Standard Clinical Care Plus Isometric Lingual Exercise (Experimental): Standard Clinical Care Plus 8-week Isometric Lingual Exercise Regimen. The isometric tongue exercises will be completed using the Madison Oral Strengthening Therapeutic (MOST) device. Baseline maximum lingual pressure will be obtained at the anterior and posterior sensors independently by gathering two sets of data (3 MOST device trials) at each site (anterior and posterior) that differ by less that 5%. During week one of the regimen, the target value of each repetition will be 60% of the maximum baseline pressure. For the remaining seven weeks of the program, the target value will be increased to 80% of the maximum. At weeks three, five, and seven, the baseline will be re-measured by phone and the 80% target value re-calculated.
  Interventions: Behavioral: Isometric Progressive Resistance Oropharyngeal Therapy

INTERVENTIONS:
Behavioral: Isometric Progressive Resistance Oropharyngeal Therapy — Tongue press exercises consist of pressing the tongue against the sensors. Isometric exercises will focus on the anterior and posterior sensor. Subjects will be given a target pressure value for both the anterior and posterior sensor locations for which to aim when doing the exercises. Visual feedback on the display will signal the subject that they have attained their target pressure goal.
  Arms: Standard Clinical Care Plus Isometric Lingual Exercise

SUMMARY:
This study is a multisite, randomized clinical trial to determine the effectiveness of an 8-week rehabilitative exercise regime performed by patients with swallowing problems, termed dysphagia, compared to a control group of patients with swallowing problems who do not exercise, but receive standard clinical care. One hundred male and female patients will take part in this study from eight participating facilities around the country.

ELIGIBILITY:
Inclusion Criteria:

* referral by a physician for swallowing evaluation because of suspected dysphagia
* complaint of difficulty swallowing
* aspiration or penetration of the laryngeal vestibule with liquids or semisolids OR post-swallow residue visible in the oral cavity, valleculae, or pharynx that is instrumentally documented by a participating SLP during a standard clinical videofluoroscopic swallowing study
* between the ages of 21 and 95
* ability to perform the exercise protocol independently or with the assistance of a caregiver
* physician approval of medical stability to participate
* decision-making capacity to provide informed consent (confirmed through discussion between the participating SLP and the subject's primary physician)

Exclusion Criteria:

* degenerative neuromuscular disease
* poorly controlled psychosis
* patient unable to complete the exercise program
* allergy to barium (used in videofluoroscopic swallowing assessment)

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Swallow Function | Baseline and 8 Weeks
  The Primary Outcome will be objectively measured from videofluoroscopic images. Improvement in swallowing is defined as a reduction in either the average Penetration/Aspiration scale score or the average Residue Scale score over the 11 swallows (3 3-ml thin liquid, 3 10-ml thin liquid, 3 3-ml semi-solid and 2 3-ml thin liquid effortful) combined with no increase in the other average score. If the series of swallows is terminated prematurely, the worst possible score (8 for Penetration/Aspiration Scale, 2 for residue) will be assigned for all uncompleted swallows.

SECONDARY OUTCOMES:
Change in Penetration/Aspiration Scale score | Baseline and Week 8
  An 8-point scale indicating occurrence, depth, clearance and patient response to material invading the laryngeal vestibule or trachea. The Penetration/Aspiration Scale score will be objectively measured from videofluoroscopic images.
Change in Residue Scale score | Baseline and Week 8
  A 3-point scale to measure post-swallow barium residue on a videofluoroscopic image. The Residue Scale score will be objectively measured from videofluoroscopic images.
Change in Bolus Transit Times | Baseline and 8 Weeks
  Durational measures of bolus flow through the oropharynx from videofluoroscopic images.
Change in Isometric Lingual Pressure | Baseline and 8 Weeks
  Maximum tongue press measured using the FDA registered Madison Oral Strenthening Therapeutic (MOST) device.
Change in Quality of Life | Baseline and 8 Weeks
  Each subject will complete a questionnaire detailing his/her quantity and variety of nutritional intake and also will complete a questionnaire (Swal-Qol) about the impact of dysphagia on his/her quality of life at baseline and week 8. It takes approximately 10 minutes to complete each questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnne Robbins, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (9):
- United States (9):
  - Northwestern University, Evanston, Illinois
  - Central Baptist Hospital, Lexington, Kentucky
  - Minneapolis Veterans Administration Health Care System, Minneapolis, Minnesota
  - Silvercrest Center for Nursing and Rehabilitation, Briarwood, New York
  - New York Hospital Queens, Flushing, New York
  - Beth Israel Medical Center, New York, New York
  - University of Pittsburgh Medical Center Passavant, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Presbyterian University Hospital, Pittsburgh, Pennsylvania
  - VA Medical Center-Memphis, Memphis, Tennessee